CLINICAL TRIAL: NCT00331955
Title: Phase I Trial of Vorinostat (NSC-701852, Suberoylanilide Hydroxamic Acid) and Doxorubicin (NSC-123127, Adriamycin)
Brief Title: Vorinostat and Doxorubicin in Treating Patients With Metastatic or Locally Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02695; MCC 14193; CDR0000471997; NCI-6970; MCC-IRB-103476; R21CA112913 (NIH); NCT00365079 (obsolete NCT alias)
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Doxorubicin; Vorinostat

ARMS (1):
- Treatment (vorinostat, doxorubicin hydrochloride) (Experimental): Patients receive oral vorinostat twice daily for 5 doses on days 1-3, 8-10, and 15-17 and doxorubicin hydrochloride IV on days 3, 10, and 17. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease after 6 courses of treatment may continue to receive vorinostat alone in the absence of disease progression.
  Interventions: Drug: doxorubicin hydrochloride; Drug: vorinostat; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of vorinostat when given together with doxorubicin in treating patients with metastatic or locally advanced solid tumors. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may help doxorubicin work better by making tumor cells more sensitive to the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of vorinostat (SAHA) and doxorubicin hydrochloride in patients with metastatic or locally advanced solid tumors.

II. Determine the maximum tolerated dose of vorinostat when administered with doxorubicin hydrochloride in patients treated with this regimen.

SECONDARY OBJECTIVES:

I. Determine the response rate (complete response [CR] and partial response [PR]) and clinical benefits rate (CR, PR, and stable disease > 12 weeks) in patients treated with this regimen.

II. Determine the pharmacokinetics and pharmacodynamics of vorinostat and doxorubicin hydrochloride and their interaction.

III. Determine the effects of vorinostat on histone acetylation in peripheral blood mononuclear cells and tumors.

IV. Determine the effects of vorinostat on DNA damage induced by doxorubicin hydrochloride as a function of topoisomerase II expression.

V. Determine the effects of vorinostat on genes and proteins crucial for the maintenance of chromatin structure.

OUTLINE: This is a non-randomized, open-label, dose-escalation study of vorinostat.

Patients receive oral vorinostat twice daily for 5 doses on days 1-3, 8-10, and 15-17 and doxorubicin hydrochloride IV on days 3, 10, and 17. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease after 6 courses of treatment may continue to receive vorinostat alone in the absence of disease progression.

Cohorts of 3-6 patients receive escalating doses of vorinostat until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to15 patients are treated at the MTD. Mandatory biopsies are required in these patients. Patients undergo blood collection and tumor biopsies periodically during the study for pharmacologic, pharmacokinetic, pharmacodynamic, and biomarker correlative studies.

After completion of study treatment, patients are followed for at least 30 days.

PROJECTED ACCRUAL: A total of 40 patients will be accrued to this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor malignancies for which no curative therapy exists
* Measurable or evaluable disease with tumor that is accessible to biopsy as determined by CT scan or ultrasound
* Skin, lymph nodes, or chest wall lesions are allowed provided measurements are confirmed by 2 independent health care professionals
* No uncontrolled CNS metastases

  * Patients with stable CNS metastases (either surgically resected, treated with gamma knife, or stable for 3 months after whole-brain radiotherapy and documented by MRI within the past 4 weeks) are eligible
* Willing to undergo pre- and post-vorinostat tumor biopsies
* Life expectancy ≥ 3 months
* ECOG performance status 0-2
* WBC > 3,000/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Hemoglobin > 9.0 g/dL
* Platelet count > 100,000/mm^3 (transfusion independent)
* Creatinine ≤ 2.0 mg/mL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 1.5 times ULN
* LVEF > 50%
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* Negative pregnancy test
* Not pregnant or nursing
* No significant active infection (e.g., pneumonia, cellulitis, or wound abscess)
* No history of cardiac failure
* No history of long QT syndrome (QTc > 470 msec)
* No history of ventricular tachycardia or fibrillation
* No history of seizures
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to vorinostat or other agents used in the study
* More than 3 weeks since prior chemotherapy or radiotherapy (2 weeks for weekly regimens)
* More than 2 weeks since prior valproic acid or any other histone deacetylase inhibitors
* No prior anthracycline exposure
* No other concurrent chemotherapy
* No concurrent hormonal therapy except for maintenance therapy with luteinizing-hormone releasing-hormone agonists
* No concurrent antiarrhythmics
* No concurrent steroids to control brain metastasis
* No concurrent colony-stimulating factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF]) during the first course of study treatment
* No other concurrent investigational agents for primary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-03; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by NCI CTCAE v3.0 | Up to 30 days after completion of treatment
Maximum tolerated dose (MTD) of vorinostat as assessed by NCI CTCAE v3.0 | 28 days

SECONDARY OUTCOMES:
Effects of vorinostat on histone acetylation | At baseline and at day 3 prior
Correlation of dose and response with biological markers for histone acetylation, Topo II expression, assays for comet moments and expression patterns of chromatin structural proteins dose | Up to 30 days after completion of study treatment
  Our initial analysis of efficacy will be descriptive and exploratory with the goal of discerning trends in various response endpoints and correlation with biological markers.
Response rate (CR and PR) and clinical benefits rate (CR, PR, and stable disease) according to RECIST | Up to 30 days after completion of study treatment
  Our initial analysis of efficacy will be descriptive and exploratory with the goal of discerning trends in various response endpoints and correlation with biological markers.
Duration of response (overall response, complete response, and stable disease) | Up to 30 days after completion of study treatment
  Using Cox regression with dose as an independent variable.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wenham, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States